CLINICAL TRIAL: NCT02063750
Title: Effectiveness of Strengthening Exercises Using the Swiss Ball for Patients With Fibromyalgia: a Randomized Controlled Trial
Brief Title: Strengthening Exercises for Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Jamil Natour, Head of Rheumatology Division, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP/UNIFESP - 1785/11
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Muscle strength exercises; Pain; Quality of life
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strengthening group (Experimental): This group perform muscle strengthening exercises using a Swiss ball of 65 cm diameter.
  Interventions: Other: strengthening exercises using a Swiss ball
- Stretching group (Active Comparator): Performed stretching exercises
  Interventions: Other: strengthening exercises

INTERVENTIONS:
Other: strengthening exercises using a Swiss ball — This group performed eight muscle strengthening exercises using a Swiss ball of 65 cm diameter and dumbbells with different loads.
  Each training session was 40 minutes long and was performed three times a week for 12 weeks. The exercises were performed in three sets of 12 repetitions, with an interval of one to two minutes of recovery between exercises, which alternated between upper limbs, lower limbs and abdomen. The load used was 60 % of one repetition maximum (1RM).
  Arms: Strengthening group
Other: strengthening exercises — The stretching group performed stretching exercises that targeted the same muscles trained in the IG. The participants remained in the stretched position for three sets of 30 s for each exercise. The total session time was 40 minutes.
  Arms: Stretching group

SUMMARY:
Objective: We evaluated the effectiveness of strengthening exercises using the Swiss ball in patients with fibromyalgia (FM).

Material and Method: Sixty FM patients were randomized into two groups: an intervention group (IG), in which patients performed muscle strength exercises using the Swiss ball, and a stretching group (SG), in which patients performed stretching exercises. All patients participated in 40-minute training sessions three times per week for 12 weeks. The IG performed the following eight strengthening exercises using a Swiss ball: lateral rise, simultaneous biceps curl, squat, two arms triceps extension, abdominal, one arm dumbbell row, reverse crucifix and crucifix. The SG performed exercises targeting the same muscle groups trained in IG. Outcome measures were as follows: visual analogue scale (VAS) for pain, 1 repetition maximum test for muscle strength; fibromyalgia impact questionnaire (FIQ) to evaluate disease impact, and short form health survey (SF-36) to assess quality of life. All participants underwent an evaluation at baseline, at 6 weeks and at 12 weeks of training. The assessor was blind to patient allocation.

ELIGIBILITY:
Inclusion Criteria:

* female with fibromyalgia according to the classification criteria of the American College of Rheumatology;
* aged between 20 and 65 years old.

Exclusion Criteria:

* uncontrolled hypertension;
* decompensated cardiac disease;
* history of syncope or exercise-induced arrhythmias and decompensated diabetes;
* severe psychiatric illness;
* history of regular exercise at least twice a week for the last 6 months;
* any other condition that could prevent the patient from performing physical exercises.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in Pain - VAS | Basline, after 6 and 12 weeks

SECONDARY OUTCOMES:
Changes in quality of life - Fibromyalgia Impact Questionnaire (FIQ) questionnaire | Baseline, after 6 and 12 weeks
Changes in muscle strength using the maximum repetition (1 RM) | Baseline, after 6 and 12 weeks
Changes in consumption of analgesics | After 6 and 12 weeks from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil